CLINICAL TRIAL: NCT02028429
Title: To Study The Proof of Concept in The Improvement of Cognition and Quality of Life in Cirrhotic Patients With Minimal Hepatic Encephalopathy by Means of a Pharmacological Intervention With Sildenafil (A Phosphodiesterase-5 Inhibitor).
Brief Title: Efficacy of Sildenafil in the Improvement of Cognition and Quality of Life in Patients With Cirrhosis of Liver. A Proof of Concept Study.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Radha K Dhiman, Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hepatology PGIMER 2012
Record Dates: First submitted 2013-12-28; First posted 2014-01-07 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Hepatic Encephalopathy.
Keywords: Minimal Hepatic Encephalopathy (MHE); Psychometric Hepatic Encephalopathy Score (PHES); Sickness Impact Profile (SIP); Model for End-stage Liver Disease (MELD); Child-Turcotte-Pugh score (CTP)
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention 'Sildenafil'. (Experimental): MHE patient receiving Sildenafil. Intervention: Sildenafil Drug Dosage: 25 mg once a day for one week followed by 25 mg twice daily for two weeks then 25 mg thrice daily for one week.
  Interventions: Drug: Sildenafil.
- 'No sildenafil' (No Intervention): Control Arm: MHE patients not receiving SIldenafil Intervention.Followed up for 4 weeks.

INTERVENTIONS:
Drug: Sildenafil. — Arm 1 :Sildenafil Drug Dosage: 25 mg once a day for one week followed by 25 mg twice daily for two weeks then 25 mg thrice daily for one week.
  Other Names: Suhagra.
  Arms: Intervention 'Sildenafil'.

SUMMARY:
The study is being conducted to evaluate the efficacy of Sildenafil (a 5-phosphodiesterase inhibitor) as a means to improve the cognitive impairment encountered in patients of minimal hepatic encephalopathy (MHE) as proposed in different studies.

This study would also assess the role of improvement of cognition as a means of improvement in quality of life.The patients will receive Sildenafil or no treatment for 4 weeks.

This study may prove and provide important therapeutic strategy for cognition impairment in patients with MHE.

DETAILED DESCRIPTION:
Primary Aim

1. To study the proof of concept in the improvement of impairment in cognition as assessed by PHES (psychometric hepatic encephalopathy score) in patients of MHE by means of pharmacological intervention by Sildenafil (a phosphodiesterase(PDE)-5 inhibitor) before and after treatment.
2. To study the impact of treatment with Sildenafil administration on the improvement in health-related quality-of-life of patients as assessed by Sickness impact profile (SIP) before and after treatment.

Secondary Aim

1. To study the impact of treatment with Sildenafil on CTP and MELD scores before and after treatment.
2. To study the impact of treatment with Sildenafil on blood ammonia and Interleukin-6 levels before and after treatment.

Study Population: The study population comprises of male adult (age 18-70 years) with cirrhosis of liver. Patients with cirrhosis of liver have been divided into two groups - with MHE and without or no MHE (NMHE) based on the test result of PHES, i.e., abnormal (MHE group) or normal (NMHE group).

Inclusion Criteria:

* Male patients aged 18-70 years diagnosed to have cirrhosis of liver at Liver Clinic of Department of Hepatology, Postgraduate Institute of Medical Education & Research(PGIMER), Chandigarh by means of clinical, biochemical and ultrasonographical/CT or liver biopsy.
* MHE will be defined by PHES ≤-5 and normal Mini-Mental State Examination (MMSE) score of ≥24.

Exclusion Criteria:

* Patients unable to give informed consent.
* H/O alcohol intake during last 12 weeks.
* Significant comorbid illness such as heart disease, respiratory disease, or renal failure.
* Any neurological disease such as Alzheimer disease, Parkinson's disease, stroke, non- hepatic metabolic encephalopathy's.
* Any anatomical deformities or disease of the penis such as Peyronie's disease.
* Patients having psychiatric illness and taking treatment with antidepressant, sedative or neuroleptics.
* Patients who start taking alcohol during the study period will be excluded.
* Patients taking vasodilators such as nitrates.
* Hepatocellular carcinoma.
* Recent history of upper GI bleed in last 6 weeks.
* Active ongoing infection.
* Electrolyte abnormality precipitating MHE.
* Color vision abnormalities.

ELIGIBILITY:
Inclusion Criteria: • Male patients aged 18-70 years diagnosed to have cirrhosis of liver at Liver Clinic of Department of Hepatology, PGIMER Chandigarh by means of clinical, biochemical and ultrasonographical/CT or liver biopsy.

* MHE will be defined by PHES ≤-5 and normal MMSE score of ≥24.

Exclusion Criteria:

* Patients unable to give informed consent.
* H/O alcohol intake during last 12 weeks.
* Significant comorbid illness such as heart disease, respiratory disease, or renal failure.
* Any neurological disease such as Alzheimer disease, Parkinson's disease, stroke, non- hepatic metabolic encephalopathy's.
* Any anatomical deformities or disease of the penis such as Peyronie's disease.
* Patients having psychiatric illness and taking treatment with antidepressant, sedative or neuroleptics.
* Patients who start taking alcohol during the study period will be excluded.
* Patients taking vasodilators such as nitrates.
* Hepatocellular carcinoma.
* Recent history of upper GI bleed in last 6 weeks.
* Active ongoing infection.
* Electrolyte abnormality precipitating MHE.
* Color vision abnormalities.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-07; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Cognition( PHES) | 4 weeks
  Improvement of impairment in cognition as assessed by PHES (Psychometric Hepatic Encephalopathy Score) in patients of MHE (Minimal hepatic Encephalopathy) by means of pharmacological intervention by sildenafil (a PDE-5 inhibitor) before and after treatment.
QOL(SIP) | 4 weeks
  To study the impact of treatment with sildenafil administration on the improvement in health-related quality-of-life of patients as assessed by sickness impact profile (SIP) before and after treatment.

SECONDARY OUTCOMES:
CTP and MELD score before and after treatment with Sildenafil. | 4 weeks
  To study the impact of treatment with sildenafil on CTP and MELD scores before and after treatment.
Blood Ammonia and Interleukin-6 levels before and after treatment with Sildenafil. | 4 weeks
  Blood Ammonia and Interleukin-6 levels before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Radha K Dhiman, MD, DM, FACG, Principal Investigator — PGIMER Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education & Research Chandigarh, Chandigarh, Chandigarh, India